CLINICAL TRIAL: NCT01397968
Title: A Phase 2 Multicenter, Double-blind, Randomized, Adjunctive, Placebo-controlled Trial With an Open-label Extension to Evaluate the Efficacy and Safety of YKP3089 in Subjects With Treatment Resistant Partial Onset Seizures
Brief Title: Efficacy and Safety of YKP3089 in Subjects With Treatment Resistant Partial Onset Seizures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YKP3089C013
Record Dates: First submitted 2011-07-18; First posted 2011-07-20 (Estimated); Results first posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Partial Epilepsy
Keywords: partial onset seizures; treatment resistant; partial epilepsy
MeSH Terms: conditions — Epilepsies, Partial | interventions — Cenobamate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- YKP3089 (Experimental)
  Interventions: Drug: YKP3089
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: YKP3089 — Capsule, dose to be titrated Tablet, dose to be titrated
  Other Names: cenobamate
  Arms: YKP3089
Drug: Placebo — Placebo capsule Placebo tablet
  Arms: Placebo

SUMMARY:
This study is to evaluate the efficacy of YKP3089 in reducing seizure frequency when compared to baseline in subjects with partial onset seizures not fully controlled despite their treatment with 1 to 3 concomitant anti-epileptic drugs.

Also to evaluate the safety and tolerability of YKP3089.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of treatment resistant partial epilepsy;
* History of epilepsy for at least 2 years;
* Have at least 3 simple partial with motor component, complex partial or secondarily generalized seizures per month with no consecutive 21 day seizure free period.
* Currently treated on a stable dose of :

  * 1 - 3 AED's for at least 12 weeks prior to randomization.
  * VNS will not be counted as AED; however the parameters must remain stable for at least 4 weeks prior to baseline.
  * Benzodiazepines taken at least once per week for epilepsy, or for anxiety or sleep disorder, will be counted as 1 AED. Therefore only a maximum of two additional approved AEDs will be allowed.

Exclusion Criteria:

1. A history of alcoholism, drug abuse, or drug addiction within the past 2 years.
2. Subject has had status epilepticus within past 1 year.
3. Subject has had greater than 2 allergic reactions to an AED or one serious hypersensitivity reaction to an AED.
4. Subjects taking felbamate with less than 18 months continuous exposure.
5. Subjects receiving phenytoin, phenobarbitone or metabolites of these drugs.
6. No active suicidal plan/intent or active suicidal thoughts in the past 6 months.
7. History of suicide attempt in the last 2 years; not more than 1 lifetime suicide attempt.
8. Subject meets criteria for current major depressive episode (within 6 months).
9. Use of intermittent rescue benzodiazepines more than once/month (1-2 doses in a 24-hour period is considered one rescue) in the one month period prior to Visit 1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2011-07-06 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2021-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Kamin, MD, Study Director — SK Life Science, Inc.
Locations (38):
- United States (16):
  - St. Joseph Hospital & Medical Center/Barrow Neurology Clinic, Phoenix, Arizona
  - Clinical Trials, Inc., Little Rock, Arkansas
  - Kaiser Permanente, Anaheim, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - Bradenton Research Center, Inc., Bradenton, Florida
  - Bluegrass Epilepsy Research, LLC, Lexington, Kentucky
  - John's Hopkins University School of Medicine, Baltimore, Maryland
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Suite 209 South, Chesterfield, Missouri
  - Ohio State University Medical Center, Columbus, Ohio
  - The University of Toledo, Toledo, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Thomas Jefferson University Comprehensive Epilepsy Center, Philadelphia, Pennsylvania
  - Neurological Clinic of Texas, P.A., Dallas, Texas
  - University of Virginia, Charlottesville, Virginia
- India (7):
  - St. Theresa's General Hospital, Hyderabad, Andhra Pradesh
  - M.S. Ramaiah Medical College and Hospital, Bangalore, Karnataka
  - Bangalore Clinisearch, Bangalore, Karnataka
  - Mallikatta Neuro Centre, Mangalore, Karnataka
  - Deenanath Mangeshkar Hospital & Research Centre, Pune, Maharashtra
  - Max Super Specialty Hospital, Saket, New Delhi
  - Nightingale Hospital, Kolkata, West Bengal
- Poland (7):
  - NZOZ Vito-Med Sp. Zo.o, Gliwice
  - NZOZ Diagnomed, Katowice
  - SPSK Nr 7 SUM w Katowicach, Gornoslaskie CM im. Prof. Leszka Gieca, Katowice
  - Malopolskie Centrum Medyczne, Krakow
  - Centrum Leczenia Padaczki i Migreny, Krakow
  - Centrum Terapii Wspolczesnej, Lodz
  - Solumed s.c., Poznan
- South Korea (8):
  - Dong-A University Medical Center, Busan
  - Keimyung University Dongsan Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Hallym University Sacred Heart Hospital, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Asan Medical Center, Seoul

REFERENCES:
- [Derived] French JA, Chung SS, Krauss GL, Lee SK, Maciejowski M, Rosenfeld WE, Sperling MR, Kamin M. Long-term safety of adjunctive cenobamate in patients with uncontrolled focal seizures: Open-label extension of a randomized clinical study. Epilepsia. 2021 Sep;62(9):2142-2150. doi: 10.1111/epi.17007. Epub 2021 Jul 13. PMID 34254673
- [Derived] Chung SS, French JA, Kowalski J, Krauss GL, Lee SK, Maciejowski M, Rosenfeld WE, Sperling MR, Mizne S, Kamin M. Randomized phase 2 study of adjunctive cenobamate in patients with uncontrolled focal seizures. Neurology. 2020 Jun 2;94(22):e2311-e2322. doi: 10.1212/WNL.0000000000009530. Epub 2020 May 14. PMID 32409485
- [Derived] Bialer M, Johannessen SI, Levy RH, Perucca E, Tomson T, White HS. Progress report on new antiepileptic drugs: a summary of the Eleventh Eilat Conference (EILAT XI). Epilepsy Res. 2013 Jan;103(1):2-30. doi: 10.1016/j.eplepsyres.2012.10.001. Epub 2012 Dec 4. PMID 23219031

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred in 4 countries (United States, Poland, Korea, India) between 06 July 2011 and 15 June 2013 when the last subject completed the double-blind period.
Pre-assignment Details: There were 285 patients screened; 63 were excluded before assignment to study group for reasons as follows:
  inclusion/exclusion criteria, withdrew by patient, other, lost to follow-up.
Groups:
- YKP3089: YKP3089: Capsule, dose to be titrated to a target dose of 200mg/day
- Placebo: Placebo: capsule, dose to be titrated to a target dose of 200mg/day
Period: Double-blind Period of Study YKP3089C013
Arm/Group | YKP3089 | Placebo
Started | 113 | 109
Completed | 102 | 99
Not Completed | 11 | 10
Period: Open-label Extension Study YKP3089C013
Arm/Group | YKP3089 | Placebo
Started (Not all subjects moved from double-blind to open-label extension.) | 76 (Not all subjects from double-blind rolled over to open-label.) | 73 (Not all subjects from double-blind rolled over to open-label.)
Completed | 40 | 37
Not Completed | 36 | 36

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | YKP3089 | Placebo | Total
Number analyzed (Participants) | 113 | 109 | 222
Age, Continuous [Median (Full Range); unit: Years] | 36 [18 to 61] | 38 [18 to 59] | 37 [18 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 51 | 109
  Male | 55 | 58 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 105 | 101 | 206
  Unknown or Not Reported | 4 | 5 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 49 | 45 | 94
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 57 | 58 | 115
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  South Korea | 22 | 19 | 41
  United States | 43 | 43 | 86
  Poland | 22 | 22 | 44
  India | 26 | 25 | 51
28-day partial-onset seizure frequency [Median (Full Range); unit: seizures/28 days] | 7.5 [0 to 187] | 5.5 [2 to 237] | 6.5 [0 to 237]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Partial-onset Seizure Frequency Per 28 Days
Description: Percent change in 28-day frequency of simple partial motor, and/or complex partial, and/or secondarily generalized tonic-clonic seizures during the 12 week treatment period relative to baseline
Time Frame: assessed per 28 days during 12 week period; change from baseline and 12 weeks reported
Measure: Median (Full Range); unit: percent seizure reduction
Arm/Group | YKP3089 | Placebo
Number analyzed (Participants) | 113 | 108
percent seizure reduction | 55.6 [-417.3 to 100.0] | 21.5 [-588.0 to 100.0]
Statistical Analysis 1: Comparison: YKP3089 vs Placebo; Test type: Superiority; p < 0.0001, Wilcoxon rank sum

2. Secondary Outcome: 50% Responder Rate
Description: Greater than or equal to 50% reduction in 28-day frequency of simple partial motor, and/or complex partial, and/or secondarily generalized tonic-clonic seizures during the 12 week treatment period relative to baseline.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | YKP3089 | Placebo
Number analyzed (Participants) | 113 | 108
Participants | 57 | 24
Statistical Analysis 1: Comparison: YKP3089 vs Placebo; Test type: Superiority; p < 0.0001, Regression, Logistic

ADVERSE EVENTS:
Time Frame: 12 week double-blind treatment period plus taper period (2-3 weeks)
Arm/Group | YKP3089 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/113 | 0/109
Serious Adverse Events (participants affected / at risk) | 3/113 | 4/109
Other Adverse Events (participants affected / at risk) | 86/113 | 69/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | YKP3089 (N=113) | Placebo (N=109)
Drug hypersensitivity reaction (Immune system disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Status epilepticus (Nervous system disorders) | 1 | 2
Convulsion (Nervous system disorders) | 0 | 1
Arteriogram coronary normal (Investigations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | YKP3089 (N=113) | Placebo (N=109)
Somnolence (Nervous system disorders) | 25 | 13
Dizziness (Nervous system disorders) | 25 | 18
Headache (Nervous system disorders) | 14 | 14
Nausea (Gastrointestinal disorders) | 13 | 5
Fatigue (General disorders) | 12 | 7
Nystagmus (Nervous system disorders) | 11 | 0
Balance disorder (Nervous system disorders) | 9 | 1
Urinary tract infection (Infections and infestations) | 9 | 2
Upper respiratory tract infection (Infections and infestations) | 8 | 5
Tremor (Nervous system disorders) | 7 | 3
Nasopharyngitis (Infections and infestations) | 7 | 1
Constipation (Gastrointestinal disorders) | 6 | 0
Diarrhea (Gastrointestinal disorders) | 6 | 0
Vomiting (Gastrointestinal disorders) | 6 | 2
Anxiety (Psychiatric disorders) | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No